CLINICAL TRIAL: NCT05157698
Title: Behavioral and Pharmacological Treatments to Enhance Weight Outcomes After Metabolic and Bariatric Surgery
Brief Title: Pharmacological and Behavioral Treatment After Bariatric Surgery
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2000029934; 1R01DK125650-01A1 (NIH)
Record Dates: First submitted 2021-11-22; First posted 2021-12-15 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Naltrexone-Bupropion combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- BWL + NB medication (Experimental): Participants randomly assigned to this arm will receive 6 months of Behavioral Weight Loss (BWL) counseling and NB medication. The naltrexone and bupropion will be taken daily in pill form.
  Interventions: Drug: Naltrexone and Bupropion Combination; Behavioral: Behavioral Weight Loss
- BWL + Placebo (Experimental): Participants randomly assigned to this arm will receive 6 months of Behavioral Weight Loss (BWL) counseling and placebo. Placebo will be inactive and taken daily in pill form.
  Interventions: Behavioral: Behavioral Weight Loss; Other: Placebo
- NB medication (Experimental): Participants randomly assigned to this arm will receive 6 months of NB medication taken daily in pill form.
  Interventions: Drug: Naltrexone and Bupropion Combination
- Placebo (Placebo Comparator): Participants randomly assigned to this arm will receive 6 months of placebo. Placebo will be inactive and taken daily in pill form.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Naltrexone and Bupropion Combination — Participants in this intervention will take active naltrexone and bupropion pills.
  Arms: BWL + NB medication; NB medication
Behavioral: Behavioral Weight Loss — Participants in this intervention will receive behavioral weight loss treatment.
  Arms: BWL + NB medication; BWL + Placebo
Other: Placebo — Participants in this intervention will take inactive (placebo) pills.
  Arms: BWL + Placebo; Placebo

SUMMARY:
This study will compare the effectiveness of behavioral and pharmacologic treatment, alone and combined, for improvements in weight loss, cardiovascular risk factors, and psychosocial functioning following metabolic and bariatric surgery.

DETAILED DESCRIPTION:
Metabolic and bariatric surgery is currently the most effective treatment for severe obesity; however, a substantial proportion of patients attain suboptimal weight losses and continue to struggle with obesity, weight regain, and related medical comorbidities after surgery. Thus, this study aims to perform a randomized double-blind placebo-controlled study to test the effectiveness of a rigorous manualized behavioral weight loss treatment and a FDA-approved weight loss agent (naltrexone+bupropion), alone and in combination, for improving weight loss, cardiovascular risk factors, and psychosocial functioning after metabolic and bariatric surgery. This study will produce important new clinical findings regarding the utility and effectiveness of pharmacotherapy and behavioral weight loss for a rapidly growing obesity subgroup and will inform care models for managing chronic and refractory obesity to enhance outcomes after metabolic and bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study (up to 18 months: 6-month treatment plus 12-month follow up)
* Have a BMI ≥30 (or BMI ≥27 with a medical comorbidity) and BMI ≤50 kg/m2
* Have had laparoscopic Roux-en-Y gastric bypass or sleeve gastrectomy
* Suboptimal weight outcomes after MBS
* Be an otherwise healthy subject without uncontrolled medical problems, as determined by the study physician and medical co-investigators (physical examination, laboratory studies).
* Have had a physical in the past year
* Read, comprehend, and write English at a sufficient level to complete study-related materials.
* For females of reproductive potential: use of highly effective contraception and agreement to use such a method during study participation
* For males of reproductive potential: use of condoms or other methods to ensure effective contraception with partner

Exclusion Criteria:

* Has a predisposition to seizures (e.g., subject with a history or evidence of seizure disorder, febrile seizures during childhood, brain tumor, cerebrovascular disease, or significant head trauma; has a family history of idiopathic seizure disorder or is currently being treated with medications or treatment regimens that lower seizure threshold).
* Has a history of anorexia nervosa or history of bulimia nervosa.
* Is currently taking a medication that is a contraindication to NB medication (e.g., MAOI, opiates).
* Is currently using other medications for weight loss.
* Has a history of allergy or sensitivity to bupropion or naltrexone.
* Has a co-existing psychiatric condition that requires hospitalization or more intensive treatment (such as bipolar mood disorders, psychotic illnesses, or severe depression)
* Has untreated hypertension with a seated systolic blood pressure > 160 mmHg, diastolic blood pressure > 100 mmHg, or heart rate > 100 beats/minute.
* Has a history of congenital heart disease, cardiovascular disease, cardiac arrhythmias requiring medication, or a history of cerebrovascular pathology including stroke.
* Has current uncontrolled hypertension.
* Has current uncontrolled Type I or Type 2 diabetes mellitus.
* Has untreated hypothyroidism with a TSH > 1.5 times the upper limit of normal for the test laboratory with repeat value that also exceeds this limit.
* Has gallbladder disease.
* Has a history of severe renal, hepatic, neurological, chronic pulmonary disease, or any other unstable medical disorder.
* Has a recent history of drug or alcohol dependence.
* Is currently in active effective treatment for eating or weight loss such as behavioral weight loss of FDA-approved weight loss medications.
* Is currently participating in another clinical study in which the subject is or will be exposed to an investigational or a non-investigational drug or device.
* Is breast-feeding or is pregnant or is not using a reliable form of birth control.
* Reports active suicidal or homicidal ideation.
* Has poor eye health

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-01-13 (Actual); Primary Completion 2027-01-12 (Estimated); Study Completion 2028-01-12 (Estimated)

PRIMARY OUTCOMES:
Change in Body Mass Index (BMI) | Baseline to after the 6-month treatment
  BMI is calculated using measured height and weight
Change in Body Mass Index (BMI) | From post-treatment (6-months) to the 12-month follow-up
  BMI is calculated using measured height and weight

SECONDARY OUTCOMES:
Change in Total cholesterol | From baseline at study enrollment to after the 6-month treatment
  Total cholesterol will be measured by bloodwork.
Change in Total cholesterol | From post-treatment (6-months) to the 12-month follow-up
  Total cholesterol will be measured by bloodwork.
Change in HbA1C | From baseline at study enrollment to after the 6-month treatment
  HbA1C will be measured by bloodwork.
  HbA1C
Change in HbA1C | From post-treatment (6-months) to the 12-month follow-up
  HbA1C will be measured by bloodwork.
  HbA1C
Change in Glucose | From baseline at study enrollment to after the 6-month treatment
  Glucose will be measured by bloodwork.
Change in Glucose | From post-treatment (6-months) to the 12-month follow-up
  Glucose will be measured by bloodwork.
Change in Loss-of-Control Eating Frequency | From baseline interview at study enrollment to after the 6-month treatment
  Loss-of-control eating frequency is a continuous variable of loss-of-control eating episodes .during the past 28 days assessed using the Eating Disorder Examination interview
Change in Loss-of-Control Eating Frequency | From post-treatment (6-months) to the 12-month follow-up
  Loss-of-control eating frequency is a continuous variable of loss-of-control eating episodes during the past 28 days assessed using the Eating Disorder Examination interview.
Change in Eating Disorder Psychopathology | From baseline interview at study enrollment to after the 6-month treatment
  Eating-disorder psychopathology is a continuous variable as assessed by the global score of the Eating Disorder Examination/Eating Disorder Examination-Questionnaire. Scores range from 0-6 (0=no eating-disorder psychopathology; 6=severe eating-disorder psychopathology).
Change in Eating Disorder Psychopathology | From post-treatment (6-months) to the 12-month follow-up
  Eating-disorder psychopathology is a continuous variable as assessed by the global score of the Eating Disorder Examination/Eating Disorder Examination-Questionnaire. Scores range from 0-6 (0=no eating-disorder psychopathology; 6=severe eating-disorder psychopathology).
Change in Food Craving | From baseline interview at study enrollment to after the 6-month treatment
  Food craving is a continuous variable of food craving as assessed by the Food Craving Inventory. Scores range from 0-5 (0=no food craving; 5=greatest food craving).
Change in Food Craving | From post-treatment (6-months) to the 12-month follow-up
  Food craving is a continuous variable of food craving as assessed by the Food Craving Inventory. Scores range from 0-5 (0=no food craving; 5=greatest food craving).
Change in Depressive Symptoms | From baseline interview at study enrollment to after the 6-month treatment
  Depressive Symptoms [ Time Frame: From baseline interview at study enrollment to after the 6-month treatment ] Depressive symptoms is a continuous variable of depressive symptomatology as assessed by the self-report measure, the Patient Health Questionnaire - 9. Total scores range from 0-27 (0=no depressive symptoms, 27=greater depressive symptoms).
  Depressive symptoms is a continuous variable of depressive symptomatology as assessed by the self-report measure, the Patient Health Questionnaire - 9. Total scores range from 0-27 (0=no depressive symptoms, 27=greater depressive symptoms).
Change in Depressive Symptoms | From post-treatment (6-months) to the 12-month follow-up
  Depressive Symptoms [ Time Frame: From baseline interview at study enrollment to after the 6-month treatment ] Depressive symptoms is a continuous variable of depressive symptomatology as assessed by the self-report measure, the Patient Health Questionnaire - 9. Total scores range from 0-27 (0=no depressive symptoms, 27=greater depressive symptoms).
  Depressive symptoms is a continuous variable of depressive symptomatology as assessed by the self-report measure, the Patient Health Questionnaire - 9. Total scores range from 0-27 (0=no depressive symptoms, 27=greater depressive symptoms).

CONTACTS AND LOCATIONS:
Overall Officials: Valentina Ivezaj, Ph.D., Principal Investigator — Yale University
Locations (1):
- Yale School of Medicine, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No